CLINICAL TRIAL: NCT06131606
Title: Effect of Stress Ball in Angiography: A Randomized Controlled Trial
Brief Title: Effect of Stress Ball in Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Dilek Güneş, Assistant Professor, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FU-SN-DG-01
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Pain, Acute
Keywords: Pain; Angiography; Anxiety; Nursing; Stress ball
MeSH Terms: conditions — Acute Pain; Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This controlled randomized study
Who Masked: Participant
Masking Description: By drawing lots, the first set was chosen to correspond to the experimental group and the second set to correspond to the control group for the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): During the angiography, the researcher asked the patient to squeeze the stress ball once for every count of three. The angiography procedure lasted approximately 25-30 minutes.
  Interventions: Behavioral: experimental group
- control group (No Intervention): No intervention other than the clinic protocol was applied to this group.

INTERVENTIONS:
Behavioral: experimental group — Patients in the experimental group were told how to use the stress ball before the procedure. The patient was then taken to the angiography unit. The stress ball was placed on the palms of the patients according to the procedure position. During the angiography, the researcher asked the patient to squeeze the stress ball once for every count of three. The angiography procedure lasted approximately 25-30 minutes. After the procedure, the NRS and STAI were filled out as a post-test 10 minutes after the patient was taken to the ward. The answers given by the patients were recorded by the researcher by marking them on the forms.
  Arms: experimental group

SUMMARY:
The target of this study was to determine the influence of stress ball application on pain and anxiety levels experienced by patients during angiography procedures.

DETAILED DESCRIPTION:
The purpose of this research was to investigate the effect of stress ball application, which is a non-pharmacologic method, on the pain and anxiety levels of patients during the angiography procedure. The present randomized controlled trial was conducted on all adult patients undergoing angiography between January 2023 and June 2023 in the Cardiovascular Surgery Clinic of a state hospital in eastern Turkey. The sample population was composed of 120 randomized patients who underwent stress ball application and received routine care. Numerical Rating Scale (NRS), Patient Information Form, and State-Trait Anxiety Inventory (STAI) were employed for data collection. The mean NRS posttest score of the experimental group patients increased significantly less than the control group (p<0.001), while the mean STAI posttest score decreased significantly (p= 0.019). A positive significant correlation was determined between the mean NRS and STAI post-test scores of the patients in the experimental group (p<0.05). It was found that the level of state-trait anxiety decreased as the pain decreased. The stress ball applied during angiography decreased the anxiety and pain levels of the patients. Stress ball application may be recommended as a complementary method to support pharmacologic treatment.

ELIGIBILITY:
Inclusion Criteria:

* no communication problems,
* being older than 18 years of age,
* having good mental health,
* undergoing wrist angiography (Radial Angiography),
* being willing to take part in the study.

Exclusion Criteria:

* Any complication during angiography.

Ages: 47 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | two weeks
  This scale, which assesses the degree of pain, aims to make the patient express their pain in numbers. It starts with no pain (0) and goes up to unbearable pain (10 or 100). The high level of pain reporting is known as a disadvantage. Miró et al. found that the validity of the NRS for pain assessment was at an acceptable level (Miró et al., 2009). Hjermstad et al. compared the Visual Analog Scale (VAS), Numerical Rating Scale (NRS), and Verbal Descriptor Scale (VDS) for the assessment of pain intensity in adults and found that the NRS was more understandable and easier to use than the VAS and VDS

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | two weeks
  The scale was developed by Spielberger et al. Its reliability and validity in our country were performed by Öner and Le Compte. The scale consists of two subunits that measure anxiety separately, but in this study, the state-trait anxiety that patients feel indirectly from the stressful situation they are in will be used. A scale of 4-point Likert-type consisting of 20-item short statements measures the state-trait anxiety level of the individual.

CONTACTS AND LOCATIONS:
Locations (1):
- Firat Universty, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yuksel D, Gunes D. The Effect of Stress Ball on Anxiety and Pain Levels in Angiography: A Randomized Controlled Trial. Cardiovasc Ther. 2024 Aug 24;2024:5049092. doi: 10.1155/2024/5049092. eCollection 2024. PMID 39742013